CLINICAL TRIAL: NCT02722356
Title: Outcomes After Implementation of a New Oxytocin Protocol for the Prevention of Postpartum Hemorrhage in Non-emergent Cesarean Sections
Brief Title: Outcomes After the Implementation of a New Oxytocin Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stacy Muir, CPT, Student Registered Nurse Anesthetist, C.R.Darnall Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 417969-1
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Complications; Cesarean Section; Adverse Reaction to Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin administered according to proposed protocol
  Interventions: Drug: Oxytocin
- Standard Practice (Active Comparator): Oxytocin administered according to standard practice at facility
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin administered per oxytocin group or standard practice group (see above)
  Other Names: Pitocin

SUMMARY:
The proposed study is a prospective, randomized, active control, open label study. One hundred sixty subjects undergoing elective cesarean section will be randomly assigned to one of two groups (n = 80 per group): the oxytocin protocol group or the standard practice group. The oxytocin protocol group will receive oxytocin boluses along with a regulated infusion according to a stepwise algorithm following delivery of the placenta. The standard practice group will receive oxytocin via a free flowing ("wide-open") infusion with a concentration of 30 IU per 500 mL of 0.9% normal saline following the delivery of the placenta. Primary outcomes include uterine tone (adequate or inadequate) as assessed by the surgeon, amount of time required to establish adequate uterine tone following the delivery of the infant, total dose of oxytocin required to establish adequate uterine tone, and total calculated blood loss based on pre-operative and post-operative hematocrit concentrations. Secondary outcomes include total estimated blood loss as agreed upon by the surgeon and the anesthesia provider, use of additional uterotonic drugs, mean arterial pressure, and incidence of oxytocin side effects (nausea, chest tightness/pain, and ST-segment changes).

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized, active control, open label between subjects design. One hundred sixty subjects will be randomly assigned to one of two groups (n = 80 per group): the oxytocin protocol group or the standard practice group. The following is a summary of the procedures used in this study:

1. All patients scheduled for an elective cesarean section will be prescreened by the investigator that is assigned as the student registered nurse anesthetist (SRNA) for that case. After obtaining informed consent and a HIPAA authorization, a full screening for eligibility will be conducted by the investigator. If determined eligible, subjects will be enrolled in the study and assigned a unique study code. Study codes will be assigned sequentially (001, 002, 003, etc.). Subjects will then be randomly allocated to one of the two groups with the use of a computer generated random number program.
2. Prior to the scheduled cesarean section investigators will record subject's age, height, weight, body mass index (BMI), parity, and gestational age. Baseline vital signs will be obtained before the start of anesthesia (blood pressure, mean arterial pressure, heart rate, respiratory rate, pulse oximetry, and temperature). A pre-operative complete blood count (CBC) will be drawn in order to obtain baseline hematocrit concentration. Procedures in this section are part of standard clinical care.
3. All subjects will have an 18-gauge IV catheter placed in the left and right upper extremity and Lactated Ringer's solution will be administered at the anesthesia provider's discretion. Standard monitors will be applied with blood pressure set to cycle at 3-minute intervals. Procedures in this section are part of standard clinical care.
4. Neuraxial anesthesia will be administered at the anesthesia provider's discretion based on patient assessment. A T4 sensory level will be established prior to beginning the cesarean section. Procedures in this section are part of standard clinical care.
5. Heart rate, ECG rhythm with ST-segment analysis, end-tidal carbon dioxide (CO2), temperature, and pulse oximetry will be monitored continuously throughout the procedure. Blood pressure and mean arterial pressure will be measured at three-minute intervals. A Foley catheter will be inserted and used to measure urine output. Procedures in this section are part of standard clinical care.
6. Throughout the procedure vasopressor drugs, crystalloids, and colloids will be administered at the anesthesia provider's discretion. Procedures in this section are part of standard clinical care.
7. Immediately after delivery of the placenta, oxytocin will be administered per the allocated group (see below). The surgeon will be blinded to the treatment group.
8. The surgeon will assess uterine tone at 3, 6, and 9 minutes following the first dose of oxytocin and deem it adequate or inadequate.
9. Subject complaints of nausea or chest tightness/pain at any time after the first dose of oxytocin will be recorded.
10. At the conclusion of the cesarean section, the amount of time required to establish adequate uterine tone following the delivery of the placenta and the total dose of oxytocin required to establish adequate uterine tone will be recorded.
11. Estimated blood loss as agreed upon by the surgeon and the anesthesia provider, need for additional uterotonic drugs, total fluid requirement (crystalloids, colloids, and blood products), total urine output, and surgical time will also be recorded at the conclusion of the procedure.
12. A post-operative CBC will be drawn 24 hours after the procedure and will be used to calculate blood loss based on the change from the pre-operative hematocrit concentration. Procedures in this section are part of standard clinical care.
13. Data will be recorded manually on a data collection sheet during the procedure and transferred to an electronic data spreadsheet. No identifying patient information will be used on data collection sheets or the electronic data spreadsheet; subjects will be identified by their unique study code.
14. Data collected will be statistically analyzed. Means, standard deviations, and covariances will be calculated for the groups. Patient characteristics such as age, weight, parity, prior cesarean section, gestational age, and baseline hematocrit will be analyzed using a multivariate analysis of variance (MANOVA) in order to determine if groups are equivalent on these parameters. An independent t-test will be used to analyze differences between the groups for continuous variables: time to adequate uterine tone, total oxytocin dose, estimated blood loss, and calculated blood loss. A Fisher's exact test will be used to analyze differences between the groups for categorical variables: uterine tone at 3, 6, and 9 minutes (adequate/inadequate), use of additional uterotonics, incidence of nausea, incidence of chest pain/tightness, and incidence of ST-segment changes. A repeated measures analysis of variance (ANOVA) with groups as the between-subjects factor and times as the within-subjects will be used to analyze differences between the groups relative to mean arterial pressure. If significance is detected, a post hoc comparison will be made using the Tukey honestly significant difference test.

Oxytocin Protocol Group Upon delivery of the placenta with confirmation from the surgeon, 3 international units (IU) of oxytocin will be administered via slow intravenous (IV) push over 30 seconds and an oxytocin infusion will be initiated at 3 IU per hour (50 mL/hr regulated by an IV pump). Investigators will wait three minutes to reassess uterine tone. If uterine tone is inadequate, an additional 3 IU bolus of oxytocin will be administered via slow IV push over 30 seconds and the oxytocin infusion will be increased to 6 IU per hour (100 mL/hr). Investigators will then wait an additional three minutes to reassess uterine tone. If uterine tone continues to be inadequate, another 3 IU bolus of oxytocin will be administered via slow IV push over 30 seconds and the oxytocin infusion will be increased to 9 IU per hour (150 mL/hr). The investigators will again wait an additional three minutes to reassess uterine tone. If uterine tone continues to be inadequate, an alternative uterotonic will be administered at the surgeon's discretion (methylergonovine 0.2 mg intramuscular [IM], carboprost tromethamine 0.25 mg IM or intramyometrial, or misoprostol 600 mcg buccal or 800-1000 mcg rectal). In the event the surgeon determines additional uterotonics are required prior to the third dose of oxytocin, the subject will be excluded from the study and additional uterotonics will be administered as necessary. Similarly, in the event the surgeon determines supplementary oxytocin is required and the protocol cannot be followed, the subject will be excluded from the study and additional oxytocin will be administered as necessary.

Standard Practice Group Upon delivery of the placenta, a free-flowing ("wide-open") oxytocin infusion will be initiated. The oxytocin infusion will be regulated at the anesthesia provider's discretion with a standard IV tubing roll-clamp and adjustments will be made as necessary after conferring with the surgeon. If adequate uterine tone is not achieved in a reasonable timeframe, the surgeon may request for an additional 20 units of oxytocin to be added to the infusion, thereby increasing the total dose of oxytocin in the 500 mL bag from 30 units to 50 units. Additional uterotonics may be requested at any time at the surgeon's discretion (methylergonovine 0.2 mg IM, carboprost tromethamine 0.25 mg IM or intramyometrial, or misoprostol 600 mcg buccal or 800-1000 mcg rectal).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with American Society of Anesthesiologists (ASA) physical status II (subjects with ASA physical status III based solely on a body mass index [BMI] ≥ 40 will be included in the study)
* Over 18 years of age
* Undergoing an elective cesarean section under neuraxial anesthesia

Exclusion Criteria:

* Maternal or obstetrician refusal
* Multiple gestation
* Ruptured membranes
* Abnormal placentation
* Preexisting coagulopathy
* Macrosomia
* Chorioamnionitis
* Diabetes mellitus (preexisting, not gestational)
* Uterine fibroids
* Contraindication to neuraxial anesthesia
* Previous allergic reaction to synthetic oxytocin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in uterine tone | 3, 6, and 9 minutes after first dose of oxytocin
  Uterine tone deemed adequate or inadequate as assessed by the surgeon
Time to adequate uterine tone | From the delivery of the infant to the completion of the cesarean section
  Amount of time (minutes) required to establish adequate uterine tone following the delivery of the infant
Oxytocin dose | Duration of cesarean section
  Total dose of oxytocin required to establish adequate uterine tone
Total calculated blood loss | 24 hours pre-op to 24 hours post-op
  Total calculated blood loss based on pre-operative and post-operative hematocrit concentrations

SECONDARY OUTCOMES:
Total estimated blood loss | Duration of cesarean section
  Total estimated blood loss as agreed upon by the surgeon and the anesthesia provider
Additional uterotonic drugs (in addition to oxytocin) required to establish adequate uterine tone: yes/no | Duration of cesarean section
Oxytocin side effects | Duration of cesarean section
  incidence of oxytocin side effects (nausea, chest tightness/pain, and ST-segment changes)

CONTACTS AND LOCATIONS:
Overall Officials: John Murphy, DNP, Study Chair — Carl R. Darnall Army Medical Center, U.S. Army Graduate Program in Anesthesia Nursing

IPD SHARING:
Plan to Share IPD: Undecided